CLINICAL TRIAL: NCT07380009
Title: Acceptability and Adherence to Different Dosing Regimens of the Multistrain Probiotic Vivomixx® 460 Neo 9 in Adults Receiving Antibiotic Therapy: a Randomized, Open-label Clinical Trial.
Brief Title: Acceptability and Adherence to Different Dosing Regimens of the Multistrain Probiotic Vivomixx® 460 Neo 9 in Adults Receiving Antibiotic Therapy.
Acronym: VIVOMIXX 460
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Thessaly (Other)
Responsible Party: Principal Investigator, Vaios Svolos, Dietitian, Postdoctoral Researcher, University of Thessaly
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 103 / 01.08.2025
Record Dates: First submitted 2025-12-21; First posted 2026-02-02 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Antibiotic Therapy
Keywords: antibiotic; probiotic; vivomixx

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- One sachet of the probiotic daily (Other): Twenty participants will receive one sachet of the probiotic daily.
  Interventions: Dietary Supplement: One sachet of the probiotic daily
- Two sachets of the probiotic daily (Other): Twenty participants will receive two sachets of the probiotic daily.
  Interventions: Dietary Supplement: Two sachets of the probiotic daily

INTERVENTIONS:
Dietary Supplement: One sachet of the probiotic daily — Twenty participants will receive one sachet of the probiotic daily.
  Arms: One sachet of the probiotic daily
Dietary Supplement: Two sachets of the probiotic daily — Twenty participants will receive two sachets of the probiotic daily.
  Arms: Two sachets of the probiotic daily

SUMMARY:
This open-label interventional study aims to evaluate the acceptability and adherence of adult participants to the multistrain probiotic Vivomixx® 460 Neo 9 when administered concurrently with antibiotic therapy. Participants are randomized to receive one of two dosing regimens: a low daily dose or a high daily dose. The study will assess the effects of these regimens on the prevention of antibiotic-associated diarrhea (AAD), gastrointestinal symptoms, and patient adherence and acceptability. The results are intended to provide evidence to optimize the clinical use of probiotics alongside antibiotics.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged over 18 years
* Initiation of oral antibiotic therapy lasting more than 3 days
* History of diarrhea during previous antibiotic treatment
* Eligible antibiotics include: (a) amoxicillin with clavulanic acid, (b) clindamycin, and (c) second- or third-generation cephalosporins
* Willingness to provide informed consent to participate in the study

Exclusion Criteria:

* Pregnancy or breastfeeding
* Age under 18 years
* Diagnosis of a chronic autoimmune disease (e.g., Crohn's disease, ulcerative colitis, rheumatoid arthritis, psoriasis)
* Diagnosis of type I or type II diabetes
* Renal or hepatic disease
* Current use of immunosuppressive medications
* Current use of other supplements, probiotics, prebiotics, or synbiotics
* Use of antibiotics within the past month
* Use of laxatives or antidiarrheal medications within the past 2 weeks
* Pre-existing diarrhea within the past 2 weeks
* Self-reported allergy to any component of the probiotic
* Psychological conditions affecting the ability to provide informed consent (e.g., dementia, psychosis, substance use)
* Gastrointestinal surgery within the past 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-12-12 (Actual); Primary Completion 2026-05-30 (Estimated); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
Adherence to the probiotic using a daily Compliance Form | From enrollment to the end of treatment at 17 days maximum
  Adherence will be assessed by recording the number of days participants took the supplement and the amount consumed, as well as by considering participant drop-out rates.
  Methods of measurement
  * Participants will be required to complete a daily Compliance Form. To minimize potential non-compliance with form completion, weekly telephone follow-up will be conducted.
  * The number of participants who complete the study and those who withdraw will be recorded.
  * When available, reasons for withdrawal will be analyzed to better understand participant responses to the intervention.
Acceptability of the probiotic supplement using an acceptability questionnaire | 2 weeks (immediately after completion of the 2-week intervention)
  Acceptability will be assessed by evaluating participants' perceptions of the intervention procedures and the administered supplement in terms of ease of use, palatability, safety, and compatibility with daily life.
  Acceptability will be measured using a structured acceptability questionnaire completed at the end of the intervention. The questionnaire will include items assessing ease of intake, difficulties in integrating the supplement into daily routines, perceived safety, overall study experience, and intention to continue product use. Responses will be recorded using a 5-point Likert scale (1 = strongly disagree to 5 = strongly agree), allowing quantitative analysis.
Daily assessment of stool type using the Bristol Stool Form Scale | From enrollment to the end of treatment at 17 days maximum
  Changes in bowel habits will be assessed by daily recording of bowel movements throughout the intervention period. Participants will document the frequency of bowel movements and stool type using the Bristol Stool Form Scale. Numbers 6,7 in the Bristol Stool Form are associated with diarrhea.

SECONDARY OUTCOMES:
Effect of the probiotic on fatigue levels | Baseline (Day 0) and 2 weeks (immediately after completion of the 2-week intervention)
  Participants will complete the Chalder Fatigue Scale (CFQ) questionnaire at the start and at the end of the intervention. Questionnaire consists of 11 Likert-scale questions designed to distinguish between physical and mental fatigue. Responses will be scored using the Likert method (0-3), yielding a total fatigue score ranging from 0 to 33, with higher scores indicating greater fatigue severity.
Effect of the intervention on participants' self-reported quality of life by WHOQOL-BREF questionnaire | Baseline (Day 0) and 2 weeks (immediately after completion of the 2-week intervention)
  Participants will complete health-related quality of life questionnaire [WHOQOL-BREF (World Health Organization Quality of Life)], which consists of 26 items rated on a 5-point Likert scale and evaluates four domains: physical health, psychological health, social relationships, and environment, along with two items assessing overall quality of life and general health. Domain scores will be calculated and transformed to a 0-100 scale according to World Health Organization guidelines, with higher scores indicating better quality of life.
Effect of the intervention on participants' self-reported quality of life by EQ-5D-5L questionnaire | Baseline (Day 0) and 2 weeks (immediately after completion of the 2-week intervention)
  Quality of life (QoL) will be assessed using EQ-5D-5L, a standardized instrument for measuring generic health status, comprising five dimensions (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression) and a Visual Analogue Scale (VAS). The EQ-5D-5L index score will be calculated using the validated country-specific value set, converting health states into a single index value ranging from 0 to 1, where higher values indicate better health-related quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: ODYSSEAS ANDROUTSOS, Principal Investigator — Lab of Clinical Nutrition and Dietetics, Department of Nutrition and Dietetics, School of Physical Education, Sports Science and Dietetics, University of Thessaly, 42100 Trikala, Greece
Locations (1):
- School of Physical Education, Sport Science and Dietetics, Trikala, Greece

IPD SHARING:
Plan to Share IPD: No